CLINICAL TRIAL: NCT06267326
Title: Case Series of Post Covid 19 Rhino Orbito Cerebral Mucormycosis in Egypt
Brief Title: World Health Organization (WHO) , COVID19 Case Series of Post Covid 19 Rhino Orbito Cerebral Mucormycosis in Egypt
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nasser Institute For Research and Treatment (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: Nasser institute
Record Dates: First submitted 2024-01-20; First posted 2024-02-20 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Mucormycosis; Rhinocerebral (Etiology); COVID-19
MeSH Terms: conditions — Mucormycosis; COVID-19 | interventions — Dosage Forms

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Twenty-one (60%) males and fourteen (40%) females, mean age was 44.17 years (Other): Twenty-one (60%) males and fourteen (40%) females, mean age was 44.17 years eighteen patients presented with COVID 19 and seventeen patients presented to our hospital post healing with history of using large doses of systemic corticosteroids. patients were managed by aggressive surgical debridement, antifungal drugs Amphotericin B and adjunctive treatment like local irrigation with amphotericin B and hyperbaric oxygen according to systemic conditions of patients. Hyperbaric oxygen was used in five patients post-surgically. all investigations were done with mean values of blood glucose level, hemoglobin and WBC were noticeably abnormal. The degree of severity, length of stay, and mortality rate were significantly correlated with the severity of systemic predisposing factors
  Interventions: Procedure: debridment
- Twenty-one (60%) males and fourteen (40%) females, mean age was 44.17 (Experimental): Twenty-one (60%) males and fourteen (40%) females, mean age was 44.17 years eighteen patients presented with COVID 19 and seventeen patients presented to our hospital post healing with history of using large doses of systemic corticosteroids. patients were managed by aggressive surgical debridement, antifungal drugs Amphotericin B and adjunctive treatment like local irrigation with amphotericin B and hyperbaric oxygen according to systemic conditions of patients. Hyperbaric oxygen was used in five patients post-surgically. all investigations were done with mean values of blood glucose level, hemoglobin and WBC were noticeably abnormal. The degree of severity, length of stay, and mortality rate were significantly correlated with the severity of systemic predisposing factors
  Interventions: Procedure: debridment

INTERVENTIONS:
Procedure: debridment — resection of dead bone
  Other Names: medication

SUMMARY:
Objectives: identify and recognize clinical Characteristics, Pathophysiology, and management of a group of patients with rhino Rhino-Orbito-Cerebral Mucormycosis infection associated with Covid 19 viral infection

ELIGIBILITY:
Inclusion Criteria:

* all patients with mucormycosis post covid 19

Exclusion Criteria:

* The patient not suffered from covid 19

Ages: 22 Years to 77 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-05-23 (Actual); Primary Completion 2022-06-12 (Actual); Study Completion 2023-08-21 (Actual)

PRIMARY OUTCOMES:
35 patients suffering from mucormycosis infection post covid 19 | 2 years
  Ratio Scale. Visual Analog Score for pain Ratio Scale. Ratio Scale. ratio scale
25 patients were cured with comorbidity and 10 pateints died | 2 years
  ordinal scale Visual Analog Score for pain
pain | two years
  Visual Analog Score for pain

SECONDARY OUTCOMES:
Visual Analog Score for pain | 2years
  pain

CONTACTS AND LOCATIONS:
Locations (1):
- Omar Elmonofy, Cairo, Egypt